CLINICAL TRIAL: NCT03565809
Title: Quality of the Management of Diabetes in Elderly People With Dementia in France. Longitudinal Study in the French National Health System Database During 2010-2015
Brief Title: Quality of the Management of Diabetes in Elderly People With Dementia in France
Acronym: DIA-FRADEM
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Collaborators: Institut National de la Santé Et de la Recherche Médicale, France (Other Government)
Responsible Party: Sponsor
Other Study IDs: RC31/16/8256
Record Dates: First submitted 2018-06-11; First posted 2018-06-21 (Actual); Last update posted 2021-09-08 (Actual); Status verified 2021-08

CONDITIONS: Alzheimer Disease
Keywords: Diabetes mellitus; Alzheimer Disease or related disorders
MeSH Terms: conditions — Alzheimer Disease; Diabetes Mellitus | interventions — Cohort Studies

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Case : ADRS group: Incidence analysis in ADRS group defined by the first recording of one of the following criteria: (i) LTD registration for ADRS (ICD-10 codes: "F00-F03", "G30", or "G31"), (ii) hospital stay reporting a diagnosis code of ADRS (similar ICD-10 codes) or (iii) reimbursement for at least one acetylcholinesterase inhibitor (rivastigmine, galantamine or donepezil) or memantine.
  Interventions: Other: Incidence analysis
- Control : non ADRS Group: Incidence analysis in non ADRS group. Each incident ADRS case was paired (1:1) to a beneficiary without any ADRS criteria, matched on age (same birth year), sex, residence area (based on of the 100 administrative 'départements') and insurance scheme.
  Interventions: Other: Incidence analysis

INTERVENTIONS:
Other: Incidence analysis — Incidence analysis between the 2 groups (ADRS/non ADRS). For each pair, an index date was defined as the ADRS identification date. In both groups, a 5-year period free of these three ADRS criteria was required before the index date, to ensure incident ADRS cases.
  Other Names: Standardized Incidence Ratios (SIR)

SUMMARY:
Along with population ageing, the association of chronic conditions such as Alzheimer's Disease and Related Syndromes (ADRS) and diabetes mellitus is increasing in clinical practice. According to ADRS severity, guidelines of diabetes care may be adapted for a personalized monitoring and treatment. The consequences on diabetes complications are not known and can also threaten dementia progression. Based on a nationwide healthcare reimbursement database, the present study aimed to compare diabetes care and the incidence of acute complications between patients with or without ADRS, in a longitudinal perspective focusing on the pivotal period of ADRS identification by the healthcare system.

ELIGIBILITY:
Inclusion Criteria:

* individuals with a first ADRS criterion in 2011 or 2012,
* prevalent diabetes mellitus, defined by a LTD with ICD-10 codes of diabetes mellitus ("E10-E14").
* at least one reimbursement in the year preceding inclusion.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Patients included in the FRADEM study : FRADEM is a nationwide case control study conducted through the French national health system database administrative data, the SNDS (systeme national des données de santé). SNDS provies reimbursement data from the entire French general population, whether subjects live at home or in a nursing home, whichever their healthcare schemes, leading to a 97% coverage of the French population in 2011.
Sampling Method: Non-Probability Sample
Enrollment: 87816 (Actual)
Dates: Start 2017-05-02 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2018-12-31 (Actual)

PRIMARY OUTCOMES:
Diabetes control | one year
  Given the absence of consensual guidelines describing the frequency of diabetes monitoring among elderly subjects, we defined a conservative minimal threshold as follows: ambulatory biological monitoring :
  * ≥ 1 annual HbA1c determination (primary endpoint)
  * ≥ 2 annual HbA1c determination
  * ≥ 1 annual lipid profile (≥ 1 annual LDL cholesterol, ≥ 1 annual triglyceride)

SECONDARY OUTCOMES:
Ocular Diabetes complications | one year
  ≥ 1 annual eye examination, defined by a visit to an ophthalmologist or a dilated fundus examination, in or out of the hospitals
Hypoglycemia | one year
  ≥ 1 annual hospitalization for hypoglycemia
ketoacidosis without coma | one year
  ≥ 1 annual hospitalization for ketoacidosis without coma
diabetic coma | one year
  - ≥ 1 annual hospitalization for diabetic coma (with ketoacidosis, hyperosmolar or hypoglycemia)
diabetic nephropathy | one year
  ≥ 1 annual hospitalization for diabetic nephropathy
diabetic neuropathy | one year
  ≥ 1 annual hospitalization for diabetic neuropathy
hospitalization for any of the 5 previous diabetes-related cause | one year
  ≥ 1 annual hospitalization for any of the 5 previous diabetes-related cause
hospitalization for falls and femoral fracture | one year
  ≥ 1 annual hospitalization for falls and femoral fracture

CONTACTS AND LOCATIONS:
Overall Officials: Virginie Gardette, MD PhD, Principal Investigator — University Hospital, Toulouse
Locations (1):
- University Hospital, Toulouse, France

REFERENCES:
- [Result] Wargny M, Gallini A, Hanaire H, Nourhashemi F, Andrieu S, Gardette V. Diabetes Care and Dementia Among Older Adults: A Nationwide 3-Year Longitudinal Study. J Am Med Dir Assoc. 2018 Jul;19(7):601-606.e2. doi: 10.1016/j.jamda.2017.12.006. Epub 2018 Feb 1. PMID 29396187